CLINICAL TRIAL: NCT05989464
Title: Self-Collected Swabs for Primary Primary Human Papilloma Virus (HPV) Screening
Brief Title: Self-Collected Swabs for Primary Human Papilloma Virus (HPV) Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Hawaii (Other)
Responsible Party: Principal Investigator, Ann Chang, Associate Professor, University of Hawaii
Other Study IDs: 2022-00672
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: HPV
Keywords: hpv; self swab; cervical cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Self-Collected Vaginal Swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Human Papilloma Virus (HPV) Self swab: Enrolled participants will be instructed to perform a self swab for genital Human Papilloma Virus (HPV) infection. Additionally, a short survey will be administered to collect demographic information, evaluate knowledge of HPV/cervical cancer, and assess acceptability of HPV self swab.
  Interventions: Diagnostic Test: Self-swab for genital HPV

INTERVENTIONS:
Diagnostic Test: Self-swab for genital HPV — Participants will insert a swab in the vagina to collect a sample for HPV testing.

SUMMARY:
In this study, the investigators will assess whether implementing a self-swab protocol for primary Human Papilloma Virus (HPV) testing is an effective method to increase cervical cancer screening in a sample of unscreened women in Hawaii. The findings of this study may support adoption of HPV self swab protocols both at Kalihi Palama Health Center (KPHC) and other Federally Qualified Health Centers (FQHC) in Hawaii.

DETAILED DESCRIPTION:
Cervical cancer is the fourth most common cancer worldwide. In the United States, the majority of cervical cancer diagnoses are made in individuals who have not been adequately screened. Cervical cancer prevention relies on adequate screening using one of three methods: pap smear cytology, Human Papilloma Virus (HPV) testing alone, or a combination of these two tests. These screening tests are performed by clinicians comfortable performing a pelvic exam, most commonly a women's health provider. Currently, less than 60% of individuals with an indication for cervical cancer screening in the Kalihi Palama Health Center (KPHC) are up-to-date on their cervical cancer screening test. Even patients who regularly see their primary care provider (PCP) can face major barriers to attending an appointment with a women's health provider. These barriers include practical issues such as inability to take time off, cost concerns, and lack of transportation. Emotional barriers include embarrassment, lack of privacy, and discomfort associated with the test.

Self-collected swabs for HPV testing is a proven strategy for populations with low screening rates. Prior studies have demonstrated increased screening rates for transgender men, African American women in the Mississippi Delta, and Women From Appalachian Ohio. Studies also reported patient evaluations of the self-sampling to be comfortable, convenient, and user-friendly; and one study found a majority preference of self-sampling over practitioner-sampling for the next screening.

Self-collected samples have also demonstrated good concordance with practitioner-collected cervical samples, as seen in multiple studies. The multiple benefits of self-swabbing without compromising screening accuracy enables the HPV self swab protocol to be an effective alternative for under screened populations. In fact, multiple countries have adopted national guidelines for self-sampled HPV screening for either under screened populations or as primary screening for all women, and more countries are piloting self-sampling to date.

In this study, the investigators will assess whether implementing a self-swab protocol for primary HPV testing is an effective method to increase cervical cancer screening in a sample of unscreened women in Hawaii. The findings of this study may support adoption of HSS protocols both at (KPHC) and other Federally Qualified Health Centers (FQHC) in Hawaii.

ELIGIBILITY:
Inclusion Criteria:

* Age of 25 years or older
* Have a cervix
* Have an indication for cervical cancer screening per Accreditation Council for Continuing Medical Education (ASCCP) guidelines
* Have been previously referred to women's health in the past 5 years or subjects have declined a women's health referral.
* Subjects must not have been seen in women's health clinic since referral was placed

Exclusion Criteria:

* Subjects unable to consent in one of the following languages: English, Chuukese, or Marshallese
* Subjects with known history of cervical cancer
* Subjects that are currently pregnant or within 3 months of giving birth

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Eligible participants will be identified by their primary care clinician at the Kalihi Palama Health Center.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of swabs with result | Within 1 week of swab collection
  Percentage of swabs with result
Percentage of participants with abnormal result | Within 1 week of swab collection
  Percentage of participants with abnormal result

SECONDARY OUTCOMES:
Self reported ease of collecting the swab | Immediately after swab is collected
  Self reported ease of collecting the swab
Willingness to collect this swab again in the future | Immediately after swab is collected
  Participants will be asked via written questionnaire: "Would you be willing to self collect this swab again in the future?"
Self reported level of worry concerning collecting self swab | Immediately after swab is collected
  Self reported level of worry concerning collecting self swab
Knowledge of HPV | Immediately after swab is collected
  Participants will be asked a true or false question concerning the prevalence of HPV in the United States on a written questionnaire.
Knowledge of cervical cancer | Immediately after swab is collected
  Participants will be asked a true or false question concerning the prevalence of cervical cancer in the United States on a written questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Chang, MD, Principal Investigator — University of Hawaii
Locations (1):
- Kalihi Palama, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No